CLINICAL TRIAL: NCT05816941
Title: The Effect of Antimicrobial Photodynamic Therapy on Periodontal Disease and Glycemic Control in Patients With Type 2 Diabetes Mellitus
Brief Title: Antimicrobial Photodynamic Therapy in Patients With Periodontal Disease and Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aPTD in Pariodontal Treatment
Record Dates: First submitted 2023-03-17; First posted 2023-04-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Periodontal Diseases; Diabetes Mellitus, Type 2; Periodontitis; Periodontal Pocket; Periodontal Attachment Loss; Periodontal Inflammation
Keywords: Type 2 Diabetes Mellitus; Periodontal Disease; Antimicrobial Photodynamic Therapy; Indocyanine Green
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2; Periodontitis; Periodontal Pocket; Periodontal Attachment Loss

STUDY DESIGN:
Intervention Model Description: Test and Control group. All patients received oral hygiene instructions followed by complete oral disinfection (removal of hard and soft deposits, scaling and root planing, mouth rinse with 0.2% chlorhexidine twice in one minute, pocket rinse with 0.2% chlorhexidine three times in ten minutes). Ultrasonic (Piezoled, KaVo) and hand instruments (Gracey curettes, Hu-Friedy, USA) were used for this purpose. Afterwards, the patients were randomly divided into test and control groups. The patients in the test group received aPDT as adjuvant treatment in pockets with PPD ≥ 5 mm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Other): Conventional Periodontal Treatment: Complete Oral Disinfection.
  Interventions: Procedure: Conventional Periodontal Treatment (Complete Oral Disinfection)
- Experimental Arm (Experimental): Conventional Periodontal Treatment (Complete Oral Disinfection) and Adjunctive Photodynamic Therapy in periodontal pockets with PPD ≥ 5 mm.
  Interventions: Procedure: Conventional Periodontal Treatment (Complete Oral Disinfection); Procedure: Adjunctive Photodynamic Therapy

INTERVENTIONS:
Procedure: Conventional Periodontal Treatment (Complete Oral Disinfection) — Oral hygiene instructions followed by complete oral disinfection (removal of hard and soft deposits, scaling and root planing, mouth rinse with 0.2% chlorhexidine twice in one minute, pocket rinse with 0.2% chlorhexidine three times in ten minutes). Ultrasonic (Piezoled, KaVo) and hand instruments (Gracey curettes, Hu-Friedy, USA) were used for this purpose.
  For the next 14 days, all patients were asked to rinse their oral cavities twice daily with 0.12% chlorhexidine.
Procedure: Adjunctive Photodynamic Therapy — Photodynamic Therapy as adjunctive treatment in pockets with PPD ≥ 5 mm. For this purpose, a Fotona XD -2 diode laser (Fotona, Ljubljana, Slovenia) with a wavelength of 810 nm, a power of 250 mW and the photosensitizing agent indocyanine green at a concentration of 1 mg/ml was used. First, the area to be irradiated was isolated, and the photosensitizing agent was applied to the periodontal pocket. After 60 seconds, the supragingival excess of the photosensitizing agent was removed by gentle rinsing with a saline solution. This was followed by irradiation for ten seconds on each side.
  For the next 14 days, all patients were asked to rinse their oral cavities twice daily with 0.12% chlorhexidine.
  Arms: Experimental Arm

SUMMARY:
Objectives: This study aimed to determine the effect of concomitant antimicrobial photodynamic therapy (aPTD) on periodontal disease and glycaemic control in patients with type 2 diabetes mellitus (T2DM).

Clinical Relevance: aPTD is a noninvasive adjunctive therapy that can positively influence the periodontal treatment outcome.

DETAILED DESCRIPTION:
Numerous studies confirm that diabetes mellitus increases the risk of gingivitis and periodontitis. However, periodontal disease also impairs glycaemic control in people with diabetes mellitus via inflammatory mediators.

Methods:

Twenty-four patients with T2DM were enrolled in the study. Periodontal tissue status and periodontal disease were assessed by measuring probing pocket depth (PPD), bleeding on probing (BOP), clinical attachment loss (CAL), plaque index (PI) and sulcus bleeding index (SBI). Glycated haemoglobin A1c (HbA1c) was measured. To determine the presence of the following periodontal pathogenic bacteria Aggregatibacter actinomycetemcomitans, Prevotella intermedia, Porphyromonas gingivalis, Tannerella forsythia and Treponema denticola, subgingival plaque samples were taken from two periodontal pockets with the greatest PPD using paper tips. Patients were randomly divided into the test and control group. In the test group, complete oral disinfection was performed in combination with aPTD. In the control group, only complete oral disinfection was performed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years
* Diabetes Mellitus type 2 with an HbA1c value > 7.0%,
* At least ten teeth in the Maxilla and Mandible
* At least four teeth with a probing pocket depth ≥ 5 mm and bleeding on probing.

Exclusion Criteria:

* Antibiotic treatment in the last four months
* Periodontal treatment in the last six months
* Any change in Antihyperglycaemic treatment three months prior to participation
* Pregnant women
* Lactating women
* Smokers
* Former smokers who had stopped smoking less than five years before participation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | At baseline
  Probing pocket depth measured using manual probe at 6 sites around each tooth. Unit: millimeters
Probing pocket depth (PPD) | 90 days after treatment
  Probing pocket depth measured using manual probe at 6 sites around each tooth. Unit: millimeters
Bleeding on probing (BOP) | At baseline
  Yes/No after probing pocket depth measurement 6 sites around each tooth. Unit: % (bleeding sites/all sites)
Bleeding on probing (BOP) | 90 days after treatment
  Yes/No after probing pocket depth measurement 6 sites around each tooth. Unit: % (bleeding sites/all sites)
Clinical attachment level (CAL) | At baseline
  This is the measurement of the position of the soft tissue attachment in relation to the cemento-enamel junction (CEJ). Two measurements are used to calculate the CAL: the probing depth and the distance from the gingival margin to the CEJ. Unit: millimeters
Clinical attachment level (CAL) | 90 days after treatment
  This is the measurement of the position of the soft tissue attachment in relation to the cemento-enamel junction (CEJ). Two measurements are used to calculate the CAL: the probing depth and the distance from the gingival margin to the CEJ. Unit: millimeters
The presence of five periodontal pathogens, Aggregatibacter actinomycetemcomitans (AA), Porphyromonas gingivalis (PG), Prevotella intermedia (PI), Tanerella forsythia (TF) and Treponema denticola (TD), | At baseline
  Plaque samples were collected with sterile paper tips after supragingival soft and hard debris had been removed according to the manufacturer's instructions. Analysis by Polymerase chain reaction (PCR) followed by hybridization against species-specific DNA probes. According to the manufacturer, the cut-off of the test is set at 10³ to 10⁴ genome equivalents
The presence of five periodontal pathogens, Aggregatibacter actinomycetemcomitans (AA), Porphyromonas gingivalis (PG), Prevotella intermedia (PI), Tanerella forsythia (TF) and Treponema denticola (TD), | 90 days after treatment
  Plaque samples were collected with sterile paper tips after supragingival soft and hard debris had been removed according to the manufacturer's instructions. Analysis by Polymerase chain reaction (PCR) followed by hybridization against species-specific DNA probes. According to the manufacturer, the cut-off of the test is set at 10³ to 10⁴ genome equivalents
HbA1c test | At baseline
  Blood sample. Unit %
HbA1c test | 90 days after treatment
  Blood sample. Unit %

SECONDARY OUTCOMES:
Plaque index (PI) | At baseline
  Yes/No at six sites around each tooth. Unit: % (sites with plaque/all sites)
Plaque index (PI) | 90 days after treatment
  Yes/No at six sites around each tooth. Unit: % (sites with plaque/all sites)
Sulcus bleeding index (SBI) | At baseline
  es/No at six sites around each tooth. Unit: % (sites with Sulcus bleeding/all sites)
Sulcus bleeding index (SBI) | 90 days after treatment
  es/No at six sites around each tooth. Unit: % (sites with Sulcus bleeding/all sites)

CONTACTS AND LOCATIONS:
Overall Officials: Rok Schara, Study Director — Assistant Professor

IPD SHARING:
Plan to Share IPD: No
All Research data will be available or shared on individual request. Example: conducting Meta-Analysis.

REFERENCES:
- [Background] Monzavi A, Chinipardaz Z, Mousavi M, Fekrazad R, Moslemi N, Azaripour A, Bagherpasand O, Chiniforush N. Antimicrobial photodynamic therapy using diode laser activated indocyanine green as an adjunct in the treatment of chronic periodontitis: A randomized clinical trial. Photodiagnosis Photodyn Ther. 2016 Jun;14:93-7. doi: 10.1016/j.pdpdt.2016.02.007. Epub 2016 Feb 24. PMID 26921460
- [Background] Braun A, Dehn C, Krause F, Jepsen S. Short-term clinical effects of adjunctive antimicrobial photodynamic therapy in periodontal treatment: a randomized clinical trial. J Clin Periodontol. 2008 Oct;35(10):877-84. doi: 10.1111/j.1600-051X.2008.01303.x. Epub 2008 Aug 17. PMID 18713259
- [Background] Lulic M, Leiggener Gorog I, Salvi GE, Ramseier CA, Mattheos N, Lang NP. One-year outcomes of repeated adjunctive photodynamic therapy during periodontal maintenance: a proof-of-principle randomized-controlled clinical trial. J Clin Periodontol. 2009 Aug;36(8):661-6. doi: 10.1111/j.1600-051X.2009.01432.x. Epub 2009 Jun 25. PMID 19563331
- [Background] Polansky R, Haas M, Heschl A, Wimmer G. Clinical effectiveness of photodynamic therapy in the treatment of periodontitis. J Clin Periodontol. 2009 Jul;36(7):575-80. doi: 10.1111/j.1600-051x.2009.01412.x. PMID 19554711
- [Background] Ge L, Shu R, Li Y, Li C, Luo L, Song Z, Xie Y, Liu D. Adjunctive effect of photodynamic therapy to scaling and root planing in the treatment of chronic periodontitis. Photomed Laser Surg. 2011 Jan;29(1):33-7. doi: 10.1089/pho.2009.2727. Epub 2010 Dec 18. PMID 21166588
- [Background] Castro Dos Santos NC, Andere NM, Araujo CF, de Marco AC, Dos Santos LM, Jardini MA, Santamaria MP. Local adjunct effect of antimicrobial photodynamic therapy for the treatment of chronic periodontitis in type 2 diabetics: split-mouth double-blind randomized controlled clinical trial. Lasers Med Sci. 2016 Nov;31(8):1633-1640. doi: 10.1007/s10103-016-2030-8. Epub 2016 Jul 22. PMID 27448223
- [Derived] Brinar S, Skvarca A, Gaspirc B, Schara R. The effect of antimicrobial photodynamic therapy on periodontal disease and glycemic control in patients with type 2 diabetes mellitus. Clin Oral Investig. 2023 Oct;27(10):6235-6244. doi: 10.1007/s00784-023-05239-0. Epub 2023 Sep 6. PMID 37672083